CLINICAL TRIAL: NCT03178422
Title: Open-Label, Multicenter Study Evaluating the Safety and Efficacy of the Nicotine Replacement Therapy Chrono Quit Smoking Solution (CQSS2) System (21mg) Compared to the NicoDerm® CQ® Patch (21mg) for Smoking Cessation in Treatment Seeking Subjects
Brief Title: Safety and Efficacy Study of the NRT CQSS2 System for Smoking Cessation in Treatment-Seeking Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chrono Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF2016-003
Record Dates: First submitted 2017-04-21; First posted 2017-06-06 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Smoking Cessation
Keywords: tobacco use cessation; smoking prevention; NRT
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: combination product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CQSS2 System (nicotine 21 mg) (Experimental): Active CQSS2 System (nicotine 21 mg) with Digital Coach. One active Drug Cartridge will be used to transdermally administer 21 mg nicotine via a 5.4% w/v solution in an aqueous EtOH mixture per day. Metered pulses of 125 µL of solution will automatically be delivered by the assembled CQSS2 (containing the Control Unit and Drug Cartridge) at Time = 0, 0.5, 1, 7, 7.5, and 13 hours.
  Interventions: Drug: CQSS2
- NicoDerm® CQ® patch (21 mg) (Active Comparator): NicoDerm® CQ® patch (21 mg) with committedquitters.com. The NicoDerm patch transdermally administers 21 mg of nicotine per day. The NicoDerm patch is applied each morning of the treatment period after waking and worn for approximately 24 hours.
  Interventions: Drug: NicoDerm CQ Patch

INTERVENTIONS:
Drug: CQSS2 — Nicotine Replacement Therapy
  Other Names: Chrono Quit Smoking Solution
  Arms: CQSS2 System (nicotine 21 mg)
Drug: NicoDerm CQ Patch — Nicotine Replacement Therapy
  Other Names: Nicotine patch
  Arms: NicoDerm® CQ® patch (21 mg)

SUMMARY:
Transdermal nicotine delivery systems are a cigarette smoking cessation aid designed to deliver nicotine into the systemic circulation via the skin. They have been found to reduce craving, thereby enhancing a patient's success for quitting smoking. However, side effects such as sleep disturbances and skin irritation, as well as incomplete smoking cessation are commonly experienced by users of such systems. Chrono Therapeutics, Inc. has developed an innovative programmable transdermal drug delivery system called the Chrono Quit Smoking Solution (CQSS2) that provides "off" periods (periods in which little to no nicotine is delivered), which is an advantage over existing systems that currently provide continuous delivery. The most important features of the CQSS2 are the periodic automatic dosing, plus the reduced side effects of sleep disturbances and potentially, skin irritation. The period when less nicotine is being delivered through the skin allows the skin an opportunity to "recover", thereby potentially reducing skin irritation. Another major benefit is the automatic dosing, which provides higher drug dosage at specific times of the day, leading to potentially greater success in quitting smoking. In this study, the CQSS2 will be used in conjunction with the Digital Coach application (app). The Digital Coach is a custom mobile app that provides behavioral support for the CQSS2. Together, the CQSS2 and the Digital Coach comprise the CQSS2 System.

DETAILED DESCRIPTION:
Study EF2016-003 is a Phase 2, randomized, two-arm, open-label, multicenter efficacy and safety study of the CQSS2 System for smoking cessation over a 6-week treatment period in healthy treatment-seeking subjects who are smokers.

PRIMARY OBJECTIVES:

To evaluate quit rates (continuous abstinence from smoking during the last 4 weeks of treatment [Visit 3 through the end of study treatment]) in smokers (more than 10 cigarettes/day) being treated with the CQSS2 System versus NicoDerm® CQ® patch

SECONDARY OBJECTIVES:

To assess the safety and tolerability of the CQSS2 System

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects must meet the following inclusion criteria:

1. Ability to participate fully in all aspects of the study.
2. Ability to understand and sign the study informed consent form.
3. English-speaking, literate males and females.
4. Age ≥18 years.
5. Smokers consuming on average >10 cigarettes per day for the past 6 months, confirmed by self report.
6. Carbon monoxide (CO) level ≥10 ppm, as determined by a Smokerlyzer breath test.
7. Subject is in good health as determined by the Investigator.
8. Subject has no known issues with completing all study visits.
9. Subject must have regular access to Verizon Wireless at home as verified by www.opensignal.com or www.sensorly.com, at home wifi, or known connectivity to Verizon Wireless.

Exclusion Criteria:

Subjects will be excluded from this study if they do not fulfill the inclusion criteria, or if any of the following conditions are observed:

1. Subjects with screening clinical laboratory tests (complete blood count [CBC] with differential and platelets, and chemistry profile) outside the normal range and considered to be clinically significant by the Investigator.
2. Subjects with severe hepatic, renal, cardiovascular, endocrine, or hematologic diseases who demonstrate abnormal electrolyte, hematology, and/or liver function (albumin, total protein, bilirubin) results on the screening blood laboratory tests, or with a history or illness that may (in the opinion of the Investigator) confound the results of the study or pose additional risk. Because these disorders may occur either alone or in combination, this judgment is left to the discretion of the Investigator caring for the subject.
3. Subjects who are immunocompromised; have an infection or suspected infection with tuberculosis (TB) or hepatitis C virus (HCV); or have a suspected infection with, or history of, human immunodeficiency virus (HIV) or hepatitis B virus (HBV).
4. Subjects with positive screening urine test for drugs of abuse, including opiates, amphetamines, barbiturates, methadone, oxycodone, benzodiazepines, cocaine, phencyclidine, methamphetamine, ecstasy, or cannabinoids; or with a history of use of cocaine, heroin, recreational drugs (e.g., MDMA/"ecstasy"), methamphetamine, or hallucinogens at any time during the past 3 months; or use of marijuana on a weekly basis for the past 3 months.
5. Subjects with recent history (past 3 months) of abuse of, or dependence on, a substance other than tobacco, including: heavy alcohol consumption (i.e., if male, drinking >4 alcoholic beverages per day for the past month and, if female, drinking >3 alcoholic beverages per day for the past month).
6. Subjects with physical examination (PE) abnormal findings considered to be clinically significant by the Investigator.
7. Subjects with tattoos that could interfere with skin assessments.
8. Subjects with any sign of infection, dermatologic disease, or condition that would inhibit transdermal absorption or might interfere with the evaluation of a test site reaction in locations where the investigational product may be used; or infection or condition (e.g., respiratory infection, strep throat) that would prevent full participation in the study.
9. Electrocardiogram (ECG) readings outside the normal range and considered to be clinically significant by the Investigator.
10. Subjects with:

    * moderately severe or severe depression, as defined by a Patient Health Questionnaire (PHQ-9) total score of ≥10, or
    * suicidal ideation, as defined by a PHQ-9 score ≥1 in response to question 9, "Thoughts that you would be better off dead, or of hurting yourself."
11. Subjects with a history of psychosis, bipolar disorder, suicide attempt, schizophrenia, or any other significant psychiatric history that the Investigator believes may interfere with the subject's participation in the study.
12. Subjects who have used an antipsychotic medication within the past 30 days. Subjects may be enrolled into the study if currently on a stable dose of antidepressant for the past 30 days and the dose is not expected to change throughout the duration of the study.
13. Subjects who require any medications that may interfere with the absorption, metabolism, or excretion of the study drug.
14. Subjects who have had a known reaction to nicotine replacement therapy (NRT) products or components.
15. Subjects who score <6 on the Visual Analogue Scale (VAS) for Motivation to Quit Smoking.
16. Women who are, or intend to become, pregnant during the course of this study, are currently breastfeeding, or women who refuse to use at least one method of birth control for the duration of the study.
17. Subjects who have used any treatments for tobacco dependence within the past 30 days.
18. Subjects who have used an investigational drug within the past 30 days or are involved in an ongoing clinical study.
19. Subjects who plan on using forms of nicotine other than cigarettes (e.g., e-cigarettes, smokeless tobacco) throughout the duration of the clinical study.
20. Subjects with a history of illness that may (in the opinion of the Investigator) confound the results of the study or pose additional risk.
21. Subjects with another household member or known relative participating in the study.
22. Subjects who have participated and been treated in any previous Chrono Therapeutics clinical study.
23. Subjects who work third shift or who otherwise stay awake all night and sleep during daylight hours.
24. Subjects who do not have access to the internet (access can be through a personal computer, smartphone, library computer, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Quit Rates for Smokers treated with the CQSS2 System vs NicoDerm CQ Patch | continuous abstinence from smoking during the last 4 weeks of treatment [Visit 3 through the end of study treatment]) in smokers (more than 10 cigarettes/day)
  Quit rates will be assessed by subject self-reporting, confirmed by Smokerlyzer testing, and documented by the Tobacco Outcome Measures Assessment. The Smoking Self Efficacy Questionnaire (SEQ12) will measure the subject's perceived ability to quit smoking.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed on an 8-point Skin Irritation Assessment scale (0 to 7) | From the time of the study drug application (6 week study period) until the last Follow-up visit.
  Any score of ≥3 will be reported as an AE

CONTACTS AND LOCATIONS:
Overall Officials: Allen Wyler, MD, Study Director — Chrono Therapeutics
Locations (5):
- United States (5):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Clinical Research Consortium, Tempe, Arizona
  - Central Kentucky Research Associates, LLC, Lexington, Kentucky
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York

IPD SHARING:
Plan to Share IPD: Undecided
Undecided